CLINICAL TRIAL: NCT05891340
Title: Effects of Prehabilitation on Postoperative Recovery in Patients Undergoing Lung Resection
Brief Title: Effects of Prehabilitation on Postoperative Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ozlem Turhan, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/2131
Record Dates: First submitted 2023-05-25; First posted 2023-06-06 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
Keywords: prehabilitation; quality of recovery; lung resection
MeSH Terms: conditions — Lung Neoplasms | interventions — Breathing Exercises

STUDY DESIGN:
Intervention Model Description: randomized, prospective
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Preoperative exercise, alcohol and smoking cessation are recommended to patients.
- Intervention (Active Comparator): Respiratory muscle exercise (two times a day) and walking (5000steps/day) are recommended to the patients preoperatively.
  Interventions: Other: Respiratory muscle exercise; Other: Endurance exercise

INTERVENTIONS:
Other: Respiratory muscle exercise — respiratory muscle exercise with inspiratory muscle trainer (two times a day)
  Arms: Intervention
Other: Endurance exercise — walking exercise 5000 steps/day
  Arms: Intervention

SUMMARY:
The study to be carried out in the Istanbul Faculty of Medicine Department of Anesthesiology was planned as a randomized, prospective study. Patients who will undergo lung resection will be included in the study.

Patients were randomized into two groups: Intervention Group includes patients who are rehabilitated preoperatively (prehabilitation), Control Group includes patients who are routinely recommended preoperative exercise, alcohol and smoking cessation. Prehabilitation consists of respiratory muscle exercise and walking is recommended to Intervention Group.

Postoperative recovery will be questioned with Quality of Recovery-15 (QoR-15) on the 2nd day and 1st month. The intensive care unit admission, postoperative pulmonary complications and length of hospital stay will be recorded.

DETAILED DESCRIPTION:
The study to be carried out in the Istanbul Faculty of Medicine Department of Anesthesiology was planned as a randomized, prospective study. Patients who will undergo lung resection will be included in the study. Patients will be informed about the study and their written consent will be obtained. Patients who do not give consent will not be included in the study.

Routine preoperative evaluation including detailed history (daily physical activity, clinical complaints at rest or exertion, if any) and physical examination will be performed on the patients. Patients were randomized into two groups: Intervention Group includes patients who are rehabilitated preoperatively (prehabilitation), Control Group includes patients who are routinely recommended preoperative exercise, alcohol and smoking cessation. Preoperative exercise, alcohol and smoking cessation are recommended to all patients. Prehabilitation consists of respiratory muscle exercise with inspiratory muscle trainer (two times a day) and walking (5000steps/day) is recommended to Intervention Group. Hospitalized patients are followed up with daily visits, and patients who are at home are followed up by phone call. All patients' induction of anesthesia and maintenance were similar.

Postoperative recovery will be questioned with Quality of Recovery-15 (QoR-15) on the 2nd day (as primary outcome) and 1st month. The duration of anesthesia, surgery duration, intensive care unit admission, postoperative pulmonary complications and length of hospital stay will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status classification system score 1-3 patients
* Patients who underwent lung resection
* Patients who agreed to participate in the study and gave written informed consent

Exclusion Criteria:

* Re-operation
* Emergency operations
* Patients with psychiatric drug use
* unability for physical exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Quality of recovery at postoperative second day | two days
  The primary aim of our study is to compare recovery of patients who have prehabilitation programme and who have not any programme by using QoR-15 questionnaire on the 2nd postoperative day.

SECONDARY OUTCOMES:
Quality of recovery at postoperative first month | one month
  Investigating recovery of patients by by using QoR-15 questionnaire
length of intensive care unit stay | two weeks
  Investigating planned or unplanned ICU admission
Length of hospital stay | one month
  patients' length of stay
Postoperative pulmonary complications | one month
  Patients' pulmonary complications such as pneumonia, atelectasis, hemorrhage, emphysema, prolonged air leak, chylothorax and respiratory failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No